CLINICAL TRIAL: NCT05169918
Title: Efficiency of Sensory Discrimination Training in Chronic Low Back Pain
Brief Title: Sensorial Discrimination in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aybike Senel, Research Assistant, PT, MSc, Research Assistant, Principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 242424
Record Dates: First submitted 2021-12-05; First posted 2021-12-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain; Back Pain; Central Sensitisation
Keywords: Chronic pain; Low back pain; Central sensitisation; Cortical reorganisation; Two point discrimination
MeSH Terms: conditions — Chronic Pain; Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: Core stabilization
- Training Group (Experimental)
  Interventions: Other: Core stabilization; Other: Sensorial Discrimination Training

INTERVENTIONS:
Other: Core stabilization — The progressive core stabilization exercise approach created by Kumar et al. will be used.
  * Stage 1; Isolation and facilitation of target muscles
  * Stage 2; Trunk stabilization training with increased load under static conditions
  * Stage 3; Development of trunk stabilization during slow controlled movement of the lumbar spine.
  * Stage 4 and 5; Lumbar stabilization during high speed and dexterous movements. The exercises will last 20-30 minutes in each sessions and twice a week for 10 weeks. The level of stage will be increased when the patients reach the aim of the stage where he/she is at. The duration of the each stage will change depending on the days the patients' need to achieve the aim of the level. For each level, at least four exercise is described.
Other: Sensorial Discrimination Training — Training group will be participate in core stabilization exercises (as describe in Control Group). Additionally, Sensorial Discrimination Training (SDT) will be applied on the low back of the patients for 20 minutes before the 20 minutes of core stabilization exercises. SDT is defined as the ability to correctly interpret the characteristics of the stimulus made to a part of the body by the patient. It aims to reverse the cortical reorganization observed in patients with chronic pain. It consists of tactile localization and graphesthesia training, which includes determining the localization and type of stimulus and recognizing the letter/number that drawn in a body part, by the patient. The training consists of five stages progressively, each stage lasting two weeks. As the participants complete the sensory tests at each stage with 90% accuracy, the next stage will be passed. If this accuracy rate is not achieved within two weeks, the stage can be extended for one week.
  Arms: Training Group

SUMMARY:
In this study, the effect of sensory discrimination training on cortical reorganization, pain and functionality in chronic nonspecific low back pain in which central sensitization is dominant will be investigated.

DETAILED DESCRIPTION:
Patients who agree to participate in the study will be assigned to Group I (core stabilization) or Group II (core stabilization+sensorial discrimination training) after being screened and randomized according to the inclusion criteria on day one. On the first day, all evaluations will be carried out by taking informed consent form from the participants. With the participants in Group I, progressive core stabilization exercises will be practiced for 20-30 minutes a day, 2 days a week for 10 weeks. In Group II, sensorial discrimination training will be studied for 20 minutes before core stabilization exercises. Core stabilization exercise will be performed in accompany with a physiotherapist who has a I. Level mat exercises certificate. At the end of each week, participants will be questioned about the use of an adjunctive intervention to treatment, including changes in medication use, or the presence of an unexpected reaction to treatment, and their responses recorded. All assessments will be repeated before treatment, at the end of the 6th week, and at the end of the 10th week. The primary outcome is cortical reorganisation which will be assessed with tactile localization, two point discrimination, pressure pain threshold. Also, proprioception of the lumbal region, lumbopelvic control, pain intensity, functionality, central sensitization, pain catastrophizing, kinesiophobia, and quality of life of the participants will be assessed. Power and Sample Size Program was used to calculate the sample size. Minimal clinically important difference (MCID) and standard deviation (SD) values were used during the calculation. For the Numerical Rating Scale, the MCID value was 4.15 and the Standard Deviation value was 3. It was calculated that a total of 15 participants, 15 participants in both groups, should be included in the study. A total of 36 participants will be included in the study by calculating a 20% probability due to the possibility of the participants being excluded from treatment or dropped out.

ELIGIBILITY:
Inclusion Criteria:

* To be between 30 and 60 years old
* To have pain lasting longer than 3 months
* To have pain intensity greater than 4 out of 10
* To have pain that is not compatible with anatomical structures and is widespread
* To get score of 40 or more from the Central Sensitization Inventory

Exclusion Criteria:

* Inability to perceive the sense of touch in the waist
* Being pregnant
* Using a pacemaker or being diagnosed with heart disease
* Having an open wound in the waist
* Using drugs that affect the central system (dopamine, etc.)
* Having a history of surgery related to the spine
* Presence of a neurological injury or disease
* Having a Body Mass Index of 30 or more
* To have a diagnosis of fibromyalgia

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Tactile localization | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  Tactile localization will be assessed as a clinical sign of cortical reorganisation. The participant will be asked to hold a pencil perpendicular to the surface at the level of the 12th thoracic vertebra in the hand ipsilateral to the tested body side (right hand if the right side of the back has been tested). The researcher will lightly touch one of the predetermined localizations and the participant will be instructed as "Use your pen to touch the point I touched as accurately as possible. Don't slide, lift the pen.". For statistical analysis, the distance between the pre-marked points and the points defined by the participant will be recorded by measuring with the caliper. This procedure will measure three times for each of the six designated points. The reliability of this test has been demonstrated in previous studies.
Two-point discrimination | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  Two-point discrimination (TPD) will be assessed as a clinical sign of cortical reorganisation. TPD is a reliable measure for detecting touch accuracy. A digital caliper (Powerfix) will be used for TPD measurements and the participant will not see the caliper during the measurement. With the participant lying prone, the researcher will measure both horizontal and vertical TPD at the L4 level bilaterally. The distance between the tips of the caliper varies between 100 mm and 5 mm, the test will be started at the maximum aperture, The distance will be reduced by 10 mm for each correct detection and increased by 5 mm for each false detection. This process will be repeated three times in descending and ascending order, and the average of the smallest distance between the caliper tips at which the participant can distinguish two separate points will be recorded as the TPD value. This measurement protocol was taken from a previous study.
Pain pressure threshold | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  Pain pressure threshold (PPT) will be assessed as a clinical sign of cortical reorganisation. Within the scope of the study, PPT measurement will be made using a digital algometer (Commander Algometer, J-Tech Medical Industries, Salt Lake City, USA). The tests will be applied to the Gluteus medius (middle and posterior part), Gluteus minimus, Gluteus maximus, Piriformis, Quadratus lumborum and Iliopsoas muscles by using a 1 cm2-pointer and increasing the pressure intensity by 1 kg/cm2 every second. The participants will be asked to tell the evaluator the point where the pressure to be applied turns into mild pain, and the average of three tests performed at 30-second intervals will be recorded in kg/cm2.

SECONDARY OUTCOMES:
Proprioception | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  Participants' sense of proprioception will be evaluated with reposition accuracy. Participants will be asked to repeat the position at three different angles, and the angle between the target position and the final movement will be recorded. The positions required from the participants is 45° lumbal flexion from the neutral position. The mean of the total value will be used as the outcome measure. Participants will be allowed to try once before the test.
Lumbopelvic motor control | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  Lumbopelvic motor control function will be evaluated using the lumbopelvic stability test described by Jung et al. In the supine position, participants will flex their hips and knees to 90° and ipsilaterally extend hips and knees to maintain abdominal pressure without touching the leg or foot on a supporting surface. Abdominal pressure will be measured with a pressurized biofeedback unit (PBU; Stabilizer, Chattanooga Group Inc., Hixson, TN). The device set to 40 mm Hg will be placed between L1 and S1 with the hip and knee flexed to 90°. The angle at which the pressure reading on the device changes during hip extension will be measured and recorded.
Pain intensity | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  Numerical Pain Scale (NAS) is a simple, reliable and short-term method that is frequently used to measure pain severity in the clinic. It is a very reliable method in the evaluation of pharmacological and non-pharmacological treatments that reduce pain. The patient is told that the most severe pain experienced is 10, and if he has no pain, the pain intensity is 0. The patient is asked to say a number between 0 and 10, which corresponds to the severity of the pain. NAS is a frequently used method in the evaluation of pain intensity in low back pain.
Central Sensitization | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  The Central Sensitization Inventory will be used to assess Central Sensitization. This questionnaire consists of 25 questions in total. The scoring of the answers to the questions is as follows: 4 points for always, 3 points for often, 2 points for sometimes, 1 point for rarely, and 0 points for never. The total score range is between 0-100 points. The cutoff score is 40. The increase in the total score indicates that the symptom grades also increase. The Turkish validity and reliability study of the questionnaire was conducted.
Pain catastrophizing | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  The level of catastrophizing the pain will be evaluated with the Pain Catastrophizing Scale (PCS). PCS is a Likert-type self-assessment scale consisting of thirteen items. Each item is evaluated between 0-4 points. The total score ranges from 0 to 52. It includes subscales of rumination, magnification, and helplessness. High scores indicate a high level of catastrophizing. The Turkish validity and reliability study was performed by İlçın N. et al.
Functionality | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  Participants' level of disability due to low back pain during activities of daily living will be evaluated with the Oswestry Low Back Pain Disability Questionnaire which consists of 10 sections that measure activities of daily living. These; pain intensity, personal care, heavy lifting, walking, sitting, standing, sleeping, sexual life, social life, travel and varying degrees of pain. Each section contains 6 questions and each section is scored between 0-5 points. The validity and reliability of the questionnaire has been demonstrated in the Turkish population.
Kinesiophobia | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  The Fear Avoidance Beliefs Questionnaire (FABQ) will be used to evaluate fear avoidance beliefs based on the effects of physical activity and work. FABQ consists of 16 questions and 2 parts. The first part of the questionnaire evaluates the attitude towards physical activities and the second part evaluates the attitude towards professional work with a 7-point Likert type scale. The physical activity section is scored between 0-24 and the labor section is scored between 0-36. The Turkish validity and reliability study of the questionnaire was conducted.
Short Form-12 | Baseline, Change from Baseline at 6th week, Change from Baseline at 10th week (end of the treatment)
  The quality of life will be assessed with Short Form-12 (SF-12). SF-12, physical functionality (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functionality (1 item), emotional role (2 items) ) and mental health (2 items) and consists of 8 sub-dimensions and 12 items. While the items related to physical and emotional role are answered as yes or no, the other items have Likert type options ranging between 3 and 6. The scores to be obtained from the physical and mental sub-dimensions range from 0 to 100, with a higher score representing better health. The Turkish validity and reliability study of the questionnaire was conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Graham A, Ryan CG, MacSween A, Alexanders J, Livadas N, Oatway S, Atkinson G, Martin DJ. Sensory discrimination training for adults with chronic musculoskeletal pain: a systematic review. Physiother Theory Pract. 2022 Sep;38(9):1107-1125. doi: 10.1080/09593985.2020.1830455. Epub 2020 Oct 20. PMID 33078667
- [Background] Kalin S, Rausch-Osthoff AK, Bauer CM. What is the effect of sensory discrimination training on chronic low back pain? A systematic review. BMC Musculoskelet Disord. 2016 Apr 2;17:143. doi: 10.1186/s12891-016-0997-8. PMID 27038609
- [Background] Ehrenbrusthoff K, Ryan CG, Gruneberg C, Martin DJ. A systematic review and meta-analysis of the reliability and validity of sensorimotor measurement instruments in people with chronic low back pain. Musculoskelet Sci Pract. 2018 Jun;35:73-83. doi: 10.1016/j.msksp.2018.02.007. Epub 2018 Mar 2. PMID 29549815